CLINICAL TRIAL: NCT06603207
Title: Causal Association Between Rheumatoid Arthritis and Periodontitis: A Mendelian Randomization Study
Brief Title: Study of the Causal Link Between Rheumatoid Arthritis and Periodontitis Using Mendelian Randomization
Acronym: RAPD-MR
Status: Not yet recruiting | Type: Observational
Sponsor: Zhibin Xu (Other)
Collaborators: Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Sponsor-Investigator, Zhibin Xu, Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Other Study IDs: KY20240918-01
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis; Periodontitis
Keywords: Mendelian Randomization; Genome-Wide Association Study (GWAS); Inflammatory Diseases; Genetic Risk Factors; SNP (Single Nucleotide Polymorphism)
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — This study uses existing GWAS data for Mendelian randomization analysis and does not involve the collection or retention of biological specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the causal relationship between rheumatoid arthritis and periodontitis using Mendelian randomization. Data will be sourced from genome-wide association studies (GWAS) to explore genetic associations and assess potential risk factors in an East Asian population.

DETAILED DESCRIPTION:
The purpose of this study is to explore the causal association between rheumatoid arthritis (RA) and periodontitis using Mendelian randomization (MR). RA and periodontitis share similar inflammatory pathways and immune responses, but their causal relationship remains unclear. This study will utilize genome-wide association studies (GWAS) data from an East Asian population to identify single nucleotide polymorphisms (SNPs) associated with RA and assess their potential impact on the risk of developing periodontitis. Statistical methods such as inverse-variance weighting, MR-Egger regression, and weighted median analysis will be employed to analyze the data. The findings may provide insights into the shared genetic basis and causal relationships between these two conditions, offering potential targets for preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Participants included in the genome-wide association study (GWAS) database.
* Subjects with available genotypic data relevant to rheumatoid arthritis and periodontitis.

Exclusion Criteria:

* Individuals without complete genotypic data or those with missing critical phenotypic information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study utilizes genetic data from an East Asian population, sourced from publicly available genome-wide association studies (GWAS) focused on rheumatoid arthritis and periodontitis.
Sampling Method: Non-Probability Sample
Enrollment: 220000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Causal Association Between Rheumatoid Arthritis and Periodontitis | Data collected from 2023 to 2024.
  This study uses Mendelian randomization to evaluate the causal relationship between rheumatoid arthritis (RA) and periodontitis in the East Asian population. The analysis utilizes genome-wide association study (GWAS) data, employing inverse variance weighting (IVW), weighted median, and MR-Egger regression methods to assess the genetic relationship and the risk contribution of RA to the development of periodontitis.

SECONDARY OUTCOMES:
Analysis of Genetic Pleiotropy and Confounders | 2023 to 2024
  Evaluation of the presence of genetic pleiotropy and its potential effect on the association between rheumatoid arthritis and periodontitis.